CLINICAL TRIAL: NCT02397447
Title: Effect of Momordica Charantia Administration on Insulin Sensitivity and Insulin Secretion in Patients With Type 2 Diabetes Mellitus, Without Pharmacological Treatment
Brief Title: Effect of Momordica Charantia Administration on Type 2 Diabetes Mellitus, Insulin Sensitivity and Insulin Secretion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Esperanza Martínez-Abundis, PhD. Esperanza Martínez-Abundis, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCHDM2
Record Dates: First submitted 2015-03-10; First posted 2015-03-25 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Momordica Charantia; Insulin secretion; Insulin sensitivity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Momordica charantia (Experimental): Two 500 mg capsules of Momordica Charantia twice daily before breakfast and dinner for 90 days
  Interventions: Drug: Momordica charantia
- Placebo (Placebo Comparator): Two 500 mg capsules of calcined magnesia twice daily before breakfast and dinner for 90 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Momordica charantia — Momordica Charantia: 2000 mg per day for three months
  Other Names: Bitter gourd, karela, balsam-pear
  Arms: Momordica charantia
Drug: Placebo — Placebo: 2000 mg per day for three months
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
The hypoglycemic effect of Momordica Charantia has been evaluated in clinical trials in patients with type 2 diabetes mellitus. Important reductions in fasting plasma glucose, glycated hemoglobin (A1C), and fructosamine were observed. It is unknown whether this improvement is due to an improvement in insulin sensitivity and insulin secretion. The purpose of this study is to evaluate the effect of the administration of Momordica Charantia on insulin sensitivity and insulin secretion in patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo controlled clinical trial is carried out in 24 patients with diagnosis of diabetes mellitus type 2 according to the criteria of the American Diabetes Association. Patients are assigned to two different arms: one group receives Momordica Charantia, 2 capsules with 500 mg twice daily before breakfast and dinner for 90 days or placebo, under the same scheme of treatment.

An oral glucose tolerance test is performed before and after the intervention. Matsuda index, Stumvoll index and Insulinogenic index are calculated to assess insulin sensitivity and insulin secretion.

Other clinical and laboratory parameters that are evaluated include: Body weight, body mass index, waist circumference, blood pressure, body fat percentage, fasting plasma glucose, A1C, creatinine, lipid profile and liver transaminases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus type 2 according to the criteria of the American Diabetes Association (<5 years), without pharmacological treatment (oral antidiabetic drugs or insulin) at least for three months before entering the study
* Fasting glucose: <210 mg/dl
* A1C: 7-9%
* Body mass index: 25-34.9 kg/m2
* Body weight without variations above or under 5% in the last three months before entering the study
* Women in childbearing years must have a contraceptive method
* Letter of consent and release signed by each patient

Exclusion Criteria:

* Pregnant or suspected pregnant women
* Woman breastfeeding
* Medications known to affect metabolism of glucose and insulin
* Personal history of liver or renal disease
* Hypertension, thyroid or cardiovascular disease decompensated
* Total cholesterol >= 240mg/dl, triglycerides >=400mg/dl, glomerular filtration rate <=60ml/min or liver transaminases >=2.5 the upper normal limit

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esperanza Martínez Abundis, PhD Science, Principal Investigator — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Momordica Charantia | Placebo
Started | 12 | 12
Completed | 10 | 10
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Momordica Charantia | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (7.3) | 47 (7.4) | 48.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 24
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24
Body weight (BW) [Mean (Standard Deviation); unit: kg] — The BW was evaluated after an overnight fast, through a bioimpedance digital scale results are reported in kilograms with a decimal.
  kg | 79.4 (9.2) | 73.6 (11.1) | 76.5 (10.4)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — The BMI was calculated by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
  kg/m^2 | 29.1 (2.4) | 28.8 (3.9) | 28.9 (3.2)
Fat mass [Mean (Standard Deviation); unit: body fat percentage] — Fat mass was measured with an electric bioimpedance scale (Model TBF-300 A; Tanita Corporation of America Inc., Arlington Heights, IL)
  body fat percentage | 36.7 (7.8) | 35.2 (8.1) | 36.0 (7.8)
Waist circumference (WC) [Mean (Standard Deviation); unit: cm] — The WC was evaluated after an overnight fast with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters
  cm | 106 (12) | 97 (11) | 101.9 (12.1)
Systolic blood pressure (SBP) [Mean (Standard Deviation); unit: mmHg] — The SBP was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of SBP. The value was expressed on mmHg.
  mmHg | 119.5 (8.9) | 116.5 (10.8) | 118.0 (9.8)
Diastolic blood pressure (DBP) [Mean (Standard Deviation); unit: mmHg] — The DBP was evaluated with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of DBP. The value was expressed on mmHg
  mmHg | 75 (4.7) | 74.2 (5.5) | 74.6 (5.0)
A1C [Mean (Standard Deviation); unit: percentage] — A liquid chromatography method was used (Bio-Rad Laboratories, Hercules, CA, USA) with an intra and inter assay coefficient of variation of 0.4% and 1.6%, respectively
  percentage | 7.8 (0.8) | 7.6 (0.6) | 7.7 (0.7)
Fasting serum glucose (FSG) [Mean (Standard Deviation); unit: mmol/L] — The glucose oxidase technique (Beckman Instruments, Inc., Brea, CA, USA) was used to determine serum glucose with an intra- and interassay coefficient of variation of<1%
  mmol/L | 8.2 (1.4) | 7.1 (1.9) | 7.6 (1.7)
2-h serum glucose [Mean (Standard Deviation); unit: mmol/L] — The glucose oxidase technique (Beckman Instruments, Inc., Brea, CA, USA) was used to determine serum glucose with an intra- and interassay coefficient of variation of<1%
  mmol/L | 17.1 (3.7) | 14.9 (4.7) | 16.0 (4.3)
AUC-glucose [Mean (Standard Deviation); unit: mmol/L/min] — The polygonal formula was used to calculate area under the curve (AUC) of glucose and insulin
  mmol/L/min | 1840 (295) | 1670 (380) | 1754.1 (344.0)
AUC-insulin [Mean (Standard Deviation); unit: pmol/L/min] — The polygonal formula was used to calculate area under the curve (AUC) of glucose and insulin
  pmol/L/min | 56562 (36078) | 41334 (22356) | 48951 (30369)
Insulinogenic index (total insulin secretion) [Mean (Standard Deviation); unit: index] — Total insulin secretion was calculated with the insulinogenic index (ΔABC insulin / ΔABC glucose)
  index | 0.29 (0.18) | 0.23 (0.14) | 0.26 (0.16)
Stumvoll index (first phase of insulin secretion) [Mean (Standard Deviation); unit: index] — First phase of insulin secretion was estimated using the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0')
  index | 557.8 (645.6) | 419.3 (769.1) | 488.6 (698.0)
Matsuda index (insulin sensitivity) [Mean (Standard Deviation); unit: index] — Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]
  index | 2.4 (1.4) | 3.8 (4.6) | 3.1 (3.4)
Total cholesterol [Mean (Standard Deviation); unit: mmol/L] — The blood sample for the determination of total cholesterol was taken after an overnight fast and was evaluated by spectrophotometry method
  mmol/L | 4.89 (0.73) | 4.41 (0.75) | 4.65 (0.76)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] — The blood sample for the determination of triglycerides was taken after an overnight fast and was evaluated by spectrophotometry method
  mmol/L | 2.31 (1.25) | 2.19 (0.76) | 2.25 (1.0)
High-density lipoprotein cholesterol (HDL-c) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for the determination of HDL-c was taken after an overnight fast and was evaluated by spectrophotometry method
  mmol/L | 1.13 (0.18) | 1.04 (0.23) | 1.09 (0.21)
Low-density lipoprotein cholesterol (LDL-c) [Median (Standard Deviation); unit: mmol/L] — The blood sample for the determination of LDL-C was taken after an overnight fast and was calculated by Friedewald formula
  mmol/L | 2.69 (0.80) | 2.35 (0.64) | 2.52 (0.73)
Very low-density lipoprotein (VLDL) [Mean (Standard Deviation); unit: mmol/L] — The blood sample for the determination of VLDL was taken after an overnight fast and was calculated as triglycerides/5
  mmol/L | 8.26 (4.48) | 7.86 (2.7) | 8.07 (3.63)
Creatinine [Mean (Standard Deviation); unit: mmol/L] — The blood sample for the determination of creatinine was taken after an overnight fast and was evaluated by spectrophotometry method
  mmol/L | 70.72 (8.84) | 61.88 (8.84) | 70.36 (8.84)
Alanine aminotransferase (ALT) [Mean (Standard Deviation); unit: U/L] — The blood sample for the determination of ALT was taken after an overnight fast and was evaluated by spectrophotometry method
  U/L | 35.4 (24.4) | 36.0 (19.7) | 35.71 (21.70)
Aspartate aminotransferase (AST) [Mean (Standard Deviation); unit: U/L] — The blood sample for the determination of AST was taken after an overnight fast and was evaluated by spectrophotometry method
  U/L | 29.0 (22.4) | 23.1 (11.3) | 26.08 (17.68)

OUTCOME MEASURES:

1. Primary Outcome: Total and First Phase of Insulin Secretion (Insulinogenic Index and Stumvoll Index) After 90 Days
Description: Total insulin secretion and first phase of insulin secretion were estimated at baseline and after 90 days using the insulinogenic index (ΔABC insulin / ΔABC glucose) and the Stumvoll index (1283+ 1.829 x insulin 30' - 138.7 x glucose 30' + 3.772 x insulin 0'), respectively
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
index
  Total insulin secretion (Insulinogenic index) | 0.41 (0.29) | 0.23 (0.12)
  First Phase of Insulin Secretion (Stumvoll index) | 1135.7 (725.0) | 309.0 (776.5)

2. Primary Outcome: Insulin Sensitivity (Matsuda Index) After 90 Days
Description: Insulin sensitivity was calculated at baseline and after 90 days with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
index | 2.1 (1.6) | 2.3 (1.0)

3. Secondary Outcome: Fasting Serum Glucose (FSG) After 90 Days
Description: The glucose oxidase technique (Beckman Instruments, Inc., Brea, CA, USA) was used to determine fasting serum glucose at baseline and after 90 days with an intra- and interassay coefficient of variation of<1
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmol/L | 7.4 (2.9) | 7.2 (2.3)

4. Secondary Outcome: A1C After 90 Days
Description: A liquid chromatography method was used to evaluate A1C at baseline and after 90 days (Bio-Rad Laboratories, Hercules, CA, USA) with an intra and inter assay coefficient of variation of 0.4% and 1.6%, respectively
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
percentage | 7.1 (1.3) | 7.1 (1.1)

5. Secondary Outcome: Total Cholesterol After 90 Days
Description: The blood sample for the determination of total cholesterol was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmol/L | 4.68 (1.02) | 4.39 (0.52)

6. Secondary Outcome: Triglycerides After 90 Days
Description: The blood sample for the determination of triglycerides was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmol/L | 1.93 (0.92) | 2.02 (0.56)

7. Secondary Outcome: High Density Lipoprotein Cholesterol (HDL-c) After 90 Days
Description: The blood sample for the determination of high density lipoprotein cholesterol was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmol/L | 1.05 (0.31) | 1.09 (0.27)

8. Secondary Outcome: Low Density Lipoprotein Cholesterol (LDL-c) After 90 Days
Description: The blood sample for the determination of low density lipoprotein cholesterol was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmol/L | 2.75 (0.96) | 2.41 (0.48)

9. Secondary Outcome: Very Low Density Lipoprotein After 90 Days
Description: The blood sample for the determination of VLDL was taken after an overnight fast and was calculated at baseline and after 90 days as triglycerides/5
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmol/L | 6.92 (3.32) | 7.22 (1.98)

10. Secondary Outcome: Alanine Aminotransferase (ALT) After 90 Days
Description: The blood sample for the determination of ALT was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
U/L | 28.1 (19.4) | 38.2 (18.9)

11. Secondary Outcome: Aspartate Aminotransferase (AST) After 90 Days
Description: The blood sample for the determination of AST was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
U/L | 23.9 (16.5) | 24.4 (6.7)

12. Secondary Outcome: Creatinine After 90 Days
Description: The blood sample for the determination of creatinine was taken after an overnight fast and was evaluated at baseline and after 90 days by spectrophotometry method
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmol/L | 70.72 (35.36) | 79.56 (0.00)

13. Secondary Outcome: Systolic Blood Pressure After 90 Days
Description: The systolic blood pressure was evaluated at baseline and after 90 days with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of SBP. The value was expressed on mmHg
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmHg | 119.6 (9.5) | 115.4 (9.8)

14. Secondary Outcome: Diastolic Blood Pressure After 90 Days
Description: The diastolic blood pressure was evaluated at baseline and after 90 days with a digital sphygmomanometer with the subject sited down on a chair after a resting period of 5 minutes on three occasions. The mean of the three measures was considered as the value of DBP. The value was expressed on mmHg
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmHg | 75.1 (6.5) | 72.6 (4.7)

15. Secondary Outcome: Body Weight (BW) After 90 Days
Description: The body weight was evaluated at baseline and after 90 days after an overnight fast, through a bioimpedance digital scale results are reported in kilograms with a decimal.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
kg | 78.0 (9.2) | 73.4 (10.8)

16. Secondary Outcome: Body Mass Index (BMI) After 90 Days
Description: The BMI was calculated at baseline and after 90 days by the square of the body height, and is universally expressed in units of kg/m^2, resulting from mass in kilograms and height in metres
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
kg/m^2 | 28.3 (1.9) | 28.9 (3.6)

17. Secondary Outcome: Fat Mass After 90 Days
Description: Fat mass was measured at baseline and after 90 days with an electric bioimpedance scale (Model TBF-300 A; Tanita Corporation of America Inc., Arlington Heights, IL)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
percentage | 36.3 (7.6) | 35.8 (6.9)

18. Secondary Outcome: Waist Circumference (WC) After 90 Days
Description: The waist circumference was evaluated at baseline and after 90 days after an overnight fast with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
cm | 104 (11) | 98 (10)

19. Secondary Outcome: 2-h Serum Glucose After 90 Days
Description: The glucose oxidase technique (Beckman Instruments, Inc., Brea, CA, USA) was used to determine serum glucose at baseline and after 90 days with an intra- and interassay coefficient of variation of<1%
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmol/L | 13.2 (4.3) | 14.3 (4.3)

20. Secondary Outcome: AUC-glucose After 90 Days
Description: The polygonal formula was used to calculate area under the curve (AUC) of glucose at baseline and after 90 days
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mmol/L/min
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
mmol/L/min | 1576 (391) | 1663 (363)

21. Secondary Outcome: AUC-insulin After 90 Days
Description: The polygonal formula was used to calculate area under the curve (AUC) of insulin at baseline and after 90 days
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: pmol/L/min
Arm/Group | Momordica Charantia | Placebo
Number analyzed (Participants) | 10 | 10
pmol/L/min | 65256 (42720) | 41310 (20292)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the 90 days of the study
Arm/Group | Momordica Charantia | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Momordica Charantia (N=12) | Placebo (N=12)
Headache (Nervous system disorders) | 4 | 3
Constipation (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Dizziness (Nervous system disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No